CLINICAL TRIAL: NCT07317310
Title: Effects of the NTU-JO Smart Program for People With Knee Osteoarthritis and Obesity: a Multicenter Pragmatic Randomized Controlled Trial
Brief Title: The NTU JO-SMART Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202509166RINB
Record Dates: First submitted 2025-12-07; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthristis; Diabetes (DM); Obesity & Overweight; Chronic Kidney Disease
Keywords: Diabetes; Chronic kidney disease; Knee osteoarthristis; obesity; Exercise; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Overweight; Renal Insufficiency, Chronic; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the intervention or control group using stratified block randomization. To ensure balance between groups regarding key prognostic factors, the randomization process will be stratified by the following variables: (1) Study center (NTUH vs. NTUH Yunlin Branch); (2) Baseline diabetes status (with T2D vs. without T2D). The allocation process will be managed through a centralized, secure web-based system. This mechanism ensures allocation concealment, preventing recruitment personnel from influencing or predicting participant assignment.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the behavioral and lifestyle intervention, it is not feasible to blind the participants or the personnel delivering the intervention (open-label design). Therefore, the primary strategy to minimize bias will be outcome assessor blinding. Research personnel responsible for conducting follow-up assessments and data collection will be distinct from those delivering the intervention and will remain blinded to the participants' group allocation throughout the study. Furthermore, the biostatisticians performing the data analysis will also be blinded to group assignment during the statistical analysis phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive a multicomponent integrated care package comprising a short-term biofeedback phase (CGM) and a long-term behavioral and exercise phase (AI-assisted exercise).
  Interventions: Behavioral: NTU-JO Smart Program
- Usual care group (No Intervention): Participants randomized to the control group will receive usual care, defined as standard clinical management for KOA and obesity provided at the outpatient departments of NTUH. This includes routine physician consultations, standard advice on weight management and physical activity, and pharmacological management as clinically indicated. No specific exercise prescription, smart equipment access, or CGM feedback will be provided.

INTERVENTIONS:
Behavioral: NTU-JO Smart Program — 1. CGM phase (weeks 1-2) During the initial 14 days of the intervention period, participants will be equipped with a CGM device. The primary goal of this short-term monitoring is to provide real-time physiological biofeedback. By visualizing the immediate fluctuations in glucose levels, participants will directly observe the impact of specific dietary choices and physical activities on their metabolic state. This "teachable moment" is designed to enhance metabolic literacy and catalyze intrinsic motivation for sustained behavioral modification.
  2. AI-assisted community-based exercise program (months 1-6) Following the initial assessment at the NTUH Exercise Counseling & Prescription Clinic, participants will engage in a 6-month, structured, multicomponent exercise program. This program integrates facility-based training using smart equipment with remote health coaching, designed to overcome common barriers to adherence in patients with KOA and obesity
  Arms: Intervention group

SUMMARY:
This study recruits patients with coexisting obesity and knee osteoarthritis (KOA) to implement the NTU-JO Smart Program, an innovative intervention integrating AI-assisted community-based exercise with continuous glucose monitoring (CGM). The primary objective is to investigate whether this intervention can improve glycemic control in this comorbid population. Other outcome measures include the risk of total knee arthroplasty (TKA), body weight changes, pain intensity scores, bone mineral density (BMD), cognitive function, as well as the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Patient-Reported Outcomes Measurement Information System (PROMIS) scores, which reflect the patients' overall functional status. The project also sought to explore the long-term association of the NTU-JO Smart Program with the development of type 2 diabetes (T2D) and major renal events, thereby facilitating patient-centered early treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 75 years.
* Obesity status: body mass index (BMI) ≥ 27 kg/m², consistent with the obesity definition defined by the Health Promotion Administration, Ministry of Health and Welfare, Taiwan.
* Diagnosis of KOA in at least one knee according to the American College of Rheumatology (ACR) criteria, with a Kellgren-Lawrence (KL) grade of 1, 2, or 3.
* Symptomatic disease: defined as a WOMAC pain subscale score (range 0-20) greater than 4 at screening.
* Sedentary lifestyle: defined as less than 30 minutes of physical activity per week for the past 6 months.
* Informed consent: willing and able to provide written informed consent and comply with all longitudinal study procedures.
* Comorbid status: participants may be included regardless of a baseline diagnosis of T2D or CKD. Stratified randomization and subgroup analyses will be conducted based on these baseline conditions.

Exclusion Criteria:

* KL grade 4 KOA in either knee.
* Diagnosis of inflammatory arthritis, such as rheumatoid arthritis or psoriatic arthritis.
* Knee arthroscopy within the past 3 months or previous surgical history of TKA.
* Recent receipt of intra-articular injections (e.g., corticosteroids, hyaluronic acid) within the past 3 months.
* Documented history of osteoporotic fracture in hospital or cloud-based medical records.
* Type 1 diabetes.
* Presence of conditions precluding safe participation in an exercise program, such as unstable cardiovascular disease or severe neurological disorders.
* Participation in another interventional clinical trial within the past 3 months.
* Engagement in dietary regimens likely to cause significant weight change (e.g., intermittent fasting, such as the 16:8 time-restricted eating) within 1 month prior to trial initiation.
* Use of any FDA-approved weight-loss medications (e.g., semaglutide, tirzepatide) within 3 months prior to trial initiation.
* History of any form of surgical treatment for weight loss.
* Current use of lithium or antipsychotics at a dose equivalent to olanzapine >20 mg/day.
* Pregnant or breastfeeding women, or women of childbearing potential without adequate contraception.
* Current malignancy (within the validity period of a catastrophic illness certificate), or any other clinical condition deemed unsuitable for participation by the investigator (investigator discretion).
* Inability to use smart devices or telecommunication tools due to severe visual/hearing impairment or lack of internet access.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2035-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with worsening glycemic control over 6 months | From enrollment to the end of intervention at 6 months
  Risk of worsening glycemic control, defined as an increase in glycated hemoglobin (HbA1c) of ≥ 0.5% from baseline assessed over the 6-month intervention period (regardless of baseline diabetes diagnosis)

SECONDARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis Index scores over 12 months | From enrollment to the end of intervention at 6 and 12 months
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function subscale score ranges from 0 to 68 (severe).
Total knee arthroplasty requirement after intervention over 12 months | From enrollment to the end of intervention over 12 months
  Incidence of progression to total knee arthroplasty requirement (defined as worsening of KL grade to grade 4 in either knee) during the follow-up period.
Change in pain intensity scores over 12 months | From enrollment to the end of intervention at 6 and 12 months
  Change in pain intensity scores on a 0-10 numeric scale.
Changes in body weight over 12 months | From enrollment to the end of intervention at 6 and 12 months
  Changes in body weight in kilograms
Change in Patient-Reported Outcomes Measurement Information System Physical Function scores over 12 months | From enrollment to the end of intervention at 6 and 12 months
  The raw Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function score is converted to a T-score centered at 50 (average), with higher T-scores meaning better ability.
Change in BMD over 24 months | From enrollment to the end of intervention at 12 and 24 months
  Change in bone mineral density assessed by dual-energy X-ray absorptiometry.
Change in Montreal Cognitive Assessment scores over 12 months | From enrollment to the end of intervention at 6 and 12 months
  The cognitive function is assessed using the Montreal Cognitive Assessment (MoCA) scores. The MoCA scores range from 0 to 30 (better).

OTHER OUTCOMES:
Number of participants with new-onset type 2 diabetes over 24 months | From enrollment to the end of intervention at 6, 12, and 24 months
  Risk of new-onset type 2 diabetes (in participants without a baseline diagnosis of diabetes), defined according to the American Diabetes Association (ADA) Standards of Care.
Number of participants with new-onset major renal events over 24 months | From enrollment to the end of intervention at 6, 12, and 24 months
  Risk of new-onset major renal events, defined as a composite endpoint: for participants without CKD at baseline, the development of new-onset CKD; or for participants with existing CKD, worsening of renal function or death (defined as a sustained decline in estimated glomerular filtration rate (eGFR) of > 40%, onset of ESRD, or death from renal causes). CKD definition: eGFR < 60 ml/min/1.73 m², or eGFR > 60 ml/min/1.73 m² accompanied by evidence of kidney damage (e.g., microalbuminuria, hematuria, or pathological findings) persisting for at least three months.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hsieh Chiang, MD, MPH, PhD, Study Chair — National Taiwan University Hospital & College of Medicine
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Taiwan
  - National Taiwan University Hospital Yunlin Branch, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: No